CLINICAL TRIAL: NCT03097783
Title: A Randomized, Multi-center, Evaluator-blinded, No-treatment Controlled Study to Evaluate the Efficacy and Safety of Restylane Perlane Lidocaine for Correction of Midface Volume Deficit and/or Midface Contour Deficiency
Brief Title: Restylane Perlane Lidocaine for Correction of Midface Volume Deficit and/or Midface Contour Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43CH1507
Record Dates: First submitted 2017-03-21; First posted 2017-03-31 (Actual); Results first posted 2021-07-21 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2021-06

CONDITIONS: Midface Volume Deficit
Keywords: hyaluronic acid, midface

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restylane Perlane Lidocaine (Experimental): Single injection and optional touch up injection with Restylane Perlane Lidocaine in Midface
  Interventions: Device: Restylane Perlane Lidocaine
- No intervention arm (No Intervention): No treatment

INTERVENTIONS:
Device: Restylane Perlane Lidocaine — Intradermal injection
  Arms: Restylane Perlane Lidocaine

SUMMARY:
This is a randomized, multi-center, evaluator-blinded, no-treatment controlled study to evaluate the efficacy and safety of Restylane Perlane Lidocaine for correction of Midface Volume Deficit and/or Midface Contour Deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Men or women aged 18 years of age or older of Chinese origin
3. Subjects willing to abstain from any other facial plastic surgical or cosmetic procedures below the level of the lower orbital rim for the duration of the study
4. Subjects seeking augmentation therapy for the midface
5. MMVS score of 2, 3 or 4 on each side of the face as assessed by the blinded evaluator

Exclusion Criteria:

1. Known/previous allergy or hypersensitivity to any injectable HA gel/local anaesthetics, e.g.lidocaine or other amide-type anaesthetics.
2. Previous surgery or tattoo in the area to be treated
3. Previous tissue augmentation therapy or contouring with any permanent (non-biodegradable) or semi-permanent filler, autologous fat, lifting threads or permanent implant below the level of the lower orbital rim.
4. Previous use of any hyaluronic acid based or collagen based biodegradable facial tissue augmentation therapy below the level of the lower orbital rim or neurotoxin within 12 months before treatment.
5. Scars or deformities, active skin disease, inflammation or related conditions, such as infection, perioral dermatitis, seborrheic eczema, rosacea, acne psoriasis and herpes zoster near or in the area to be treated.
6. Other condition preventing the subject from entering the study in the Investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Med AB, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Wu Y, Li B, Mu X, Li L. Lifting the midface using a hyaluronic acid filler with lidocaine: A randomized multi-center study in a Chinese population. J Cosmet Dermatol. 2022 Dec;21(12):6710-6716. doi: 10.1111/jocd.15286. Epub 2022 Oct 25. PMID 35925834

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restylane Perlane Lidocaine | No Intervention Arm
Started | 132 | 37
Completed | 123 | 31
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restylane Perlane Lidocaine | No Intervention Arm | Total
Number analyzed (Participants) | 132 | 37 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 132 | 36 | 168
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (10.3) | 48 (11.1) | 46 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 35 | 154
  Male | 13 | 2 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 132 | 37 | 169
Region of Enrollment [Number; unit: participants]
  China | 132 | 37 | 169

OUTCOME MEASURES:

1. Primary Outcome: Percent Responders With 1 Point Improvement on the Medicis Midface Volume Scale
Description: The primary objective is to demonstrate superiority of Perlane-Lido relative to no-treatment in the treatment of Midface volume Deficit and/or Midface Contour Deficiency by comparing the percent responders, defined by at least 1 point improvement from baseline on the MMVS on both sides of the face, as measured by blinded evaluator at 6 months.
  Medicis Midface Volume Scale (MMVS) is a 4-grade scale assesses the fullness of the midface from Fairly Full (1) to Substantial Loss of Fullness (4) as described below. The blinded evaluator and treating investigator will rate the subject's right and left midface for severity of volume deficiency using the MMVS at all applicable study visits.
  1. Fairly full midface
  2. Mild loss of fullness in midface area
  3. Moderate loss of fullness with slight hollowing below malar prominence
  4. Substantial loss of fullness in the midface area, clearly apparent hollowing below malar prominence
Time Frame: 6 month
Population: All summaries will be done separately for Group A and B. For statistical inference,only Group B will be used.
Measure: Count of Participants; unit: Participants
Arm/Group | Restylane Perlane Lidocaine | No Intervention Arm
Number analyzed (Participants) | 110 | 37
Participants | 67 | 8

ADVERSE EVENTS:
Time Frame: 1 year.
Description: The question asked will be "Since your last clinical visit have you had any health problems?" Information on AEs can also be obtained from signs and symptoms detected during each examination or from a laboratory test, observations by the study personnel, subject diaries or spontaneous reports from the subjects.
Arm/Group | Restylane Perlane Lidocaine | No Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/37
Other Adverse Events (participants affected / at risk) | 0/110 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT03097783/Prot_002.pdf
  • Statistical Analysis Plan (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/83/NCT03097783/SAP_003.pdf